CLINICAL TRIAL: NCT06766435
Title: Evaluation of the Abbott i-STAT TBI Biomarker Test for Effect on Decreasing CT Utilization Among Adult Emergency Department Patients With Suspected Traumatic Brain Injury
Brief Title: Evaluation of the Abbott i-STAT TBI Biomarker Test
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Abbott Point of Care (Industry)
Responsible Party: Principal Investigator, Shameeke Taylor, Assistant Professor of Emergency Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY-24-01057; CRS-2024-001-257 (Other Grant/Funding Number: Abbott Point of Care)
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury
Keywords: Point of Care Testing; Emergency Care; Clinical Decision Making; Head Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma

STUDY DESIGN:
Intervention Model Description: Multisite randomized controlled clinical trial
Masking Description: Patient is randomized to the intervention or control arm after consent is obtained. There is no masking for the treatment arm assignment. In the non-notification arm (control arm) participants and care providers will not learn the results of the i-STAT TBI test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Notification Arm (Abbott iSTAT TBI test) (Experimental): The ED clinicians caring for the enrolled patient, along with the patient, receive the TBI blood test result with just-in-time education on the TBI test to aid in clinical decision making.
  Interventions: Device: i-STAT TBI Test
- Non-Notification Arm (Control) (No Intervention): Clinicians and enrolled patients do not receive the TBI blood test result.

INTERVENTIONS:
Device: i-STAT TBI Test — The Abbott i-STAT TBI test result is shared with the enrolled patient and treating clinicians.
  Other Names: Abbott iSTAT Alinity
  Arms: Notification Arm (Abbott iSTAT TBI test)

SUMMARY:
According to the Centers for Disease Control and Prevention, approximately 200,000 hospitalizations occurred in 2020 related to Traumatic Brain Injury (TBI), which does not include many TBIs treated only in emergency departments, urgent care, primary care, or that are not evaluated by a clinician. Head CT is a critical component of care for severe TBI, however in mild TBI there is practice variation with a wider risk to benefit estimation for obtaining head CT imaging. Potential disadvantages of head CT include longer Emergency Department (ED) length of stay (LOS), higher costs, and diagnostic radiation exposure. The i-STAT TBI test is a panel of in vitro diagnostic immunoassays for the quantitative measurements of glial fibrillary acidic protein (GFAP) and ubiquitin carboxyl-terminal hydrolase L1 (UCH-L1) in whole blood and a semi-quantitative interpretation of test results derived from these measurements, using the i-STAT Alinity instrument. This biomarker test is cleared for use in adults with mild TBI (Glasgow Coma Scale 13-15) within 24 hours of injury, to aid in determining the need for head CT imaging. Currently, CT head imaging for adults with suspected mild TBI is obtained based on clinicians' usual practice patterns and beliefs about patient expectations. Prior research has demonstrated the blood TBI test may reduce unnecessary CT scans by up to 40%, however the impact on head CT ordering has not yet been studied prospectively. It is important to understand the extent to which a negative TBI biomarker result empowers a clinician to cancel a previously ordered head CT. Given that adult patients with mild TBI often present to EDs, which have access to CT scanners, this is a key setting to assess real-world impact of the i-STAT TBI test on CT head utilization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Head injury within 24 hours of research blood collection
* CT head ordered as part of routine care, not yet completed.
* Glasgow Coma Scale (GCS) 13 - 15

Exclusion Criteria:

* Unknown whether head injury occurred, and signs of head injury are absent
* Previously enrolled in this study in the past 30 days
* Prisoner or in police custody or known pregnancy
* Suspected current ischemic or hemorrhagic stroke
* Suspected open or depressed skull fracture, or signs of skull base fracture
* History of multiple sclerosis
* Venipuncture not feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of Head CT scans canceled | Within 24 hours of Traumatic Brain Injury
  Number of head CTs canceled in patients not on anticoagulants as measurement of percentage of reduction in the number of canceled head CTs out of total head CTs ordered (total number and percentage)

SECONDARY OUTCOMES:
Subset of Number of Head CT scans completed | Within 24 hours of Traumatic Brain Injury
  If the i-STAT TBI test results had been strictly adhered to by clinicians, subset of negative i-STAT TBI test results, Potential reduction in the number of completed head CTs (canceled) out of total head CTs ordered (total number and percentage)
ED Length of Stay | Day 1 after patient ED care visit has ended
  Length of stay for the Emergency Department patient encounter
Number of cancellations of head CT scan order in patients on anticoagulants | Day 1 after patient ED care visit has ended
  Number of cancellations in head CTs in patients on anticoagulation
Patient Satisfaction Scale | At 14 days after ED visit
  Assessment of patient satisfaction with care during ED visit. Full scale from 1 (worst care possible) to 10 (best care possible)
Number of head CT scans completed | At 14 days after ED visit
  Number of head CT scans completed for patients within 14 days after index ED visit
Stress of Uncertainty Scale (SUS) | Day 1 during patient ED care visit
  Clinicians vary in their use of diagnostic testing and treatments, and stress of uncertainty may be one explanation for this variation. The stress of uncertainty scale measures clinician tolerance of uncertainty during patient care. SUS scores range from 15-90 with a higher score indicating greater fear of uncertainty.
Malpractice Fear Scale (MFS) Scores | Day 1 during patient ED care visit
  Malpractice Fear Scale (MFS) scores. MFS scores range from 6 to 36 with a higher score indicating greater fear of malpractice.
Whole blood concentrations of GFAP (glial fibrillary acidic protein) | Day 1 during patient ED care visit
  Whole blood concentrations for GFAP on the iSTAT device. Biomarker for use with mild TBI within 24 hours of injury to aid in determining the need for head CT imaging.
Whole blood concentrations of UCH-L1 (ubiquitin C-terminal hydrolase L1) | Day 1 during patient ED care visit
  Whole blood concentrations for UCH-L1 on the iSTAT device. Biomarker for use with mild TBI within 24 hours of injury to aid in determining the need for head CT imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Shameeke Taylor, MD, MPH, MSCR, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Mount Sinai Morningside, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Mount Sinai West, New York, New York

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time.